CLINICAL TRIAL: NCT01948427
Title: Long-Term Registry of Patients With Urea Cycle Disorders (UCDs)
Brief Title: Observational Study That Will Collect Information on Patients With Urea Cycle Disorders (UCDs)
Acronym: THRIVE
Status: Terminated | Type: Observational
Why Stopped: the study was terminated due to the primary end point being met.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: HPN-100-014
Record Dates: First submitted 2013-09-16; First posted 2013-09-23 (Estimated); Results first posted 2021-02-18 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Urea Cycle Disorder
Keywords: UCD; BUPHENYL; RAVICTI; Urea; Urea cycle disorder; Glycerol phenylbutyrate; Benzoate; Sodium phenylbutyrate; Ornithine transcarbamylase (OTC); Argininosuccinate synthetase (ASS); Argininosuccinate lyase (ASL); Carbamyl phosphate synthetase (CPS); Arginine; Citrulline; Ammonia
MeSH Terms: conditions — Urea Cycle Disorders, Inborn; Ornithine Carbamoyltransferase Deficiency Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
THRIVE is an observational study that will collect information on patients with UCDs. THRIVE will follow enrolled participants for up to 10 years. As an observational study, enrolled patients will not be required to make any additional office visits or take any medicine outside of normal care.

DETAILED DESCRIPTION:
UCDs disproportionately affect children and females: depending on the severity of the defect, a UCD can manifest shortly after birth or later in life. This study will track long-term outcomes in UCD patients and effects of ammonia-scavenging agents on neuropsychological functions of UCD patients.

This is a non-interventional, multi-center registry to be conducted in patients with UCDs. Investigators will prescribe treatments based on usual clinical practice, and there will be no restrictions on the use of commercially available medications. As an observational study, this study will not change the patient/ healthcare provider relationship, nor influence the healthcare provider's drug prescription or the therapeutic management of the patient.

Patients with UCDs will be recruited and invited to attend a Baseline visit. After eligible patients are enrolled, retrospective and baseline data will be collected. Patients will be followed for up to 10 years, during which time they will be assessed by their healthcare provider. Patients and healthcare provider will be asked to report episodes of hyperammonemic crisis, available ammonia values, and other information.

Study acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed or suspected diagnosis of UCD
* Signed informed consent/Health Insurance Portability and Accountability Act (HIPAA) Authorization and medical records release

Exclusion Criteria:

* Any other reason that, in the Investigator's opinion, makes the patient unsuitable to participate in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a confirmed or suspected diagnosis of UCD
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2013-09-25 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- United BioSource Corporation, Blue Bell, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: THRIVE Registry Website — https://www.thriveregistry.com/index.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Sodium Phenylbutyrate: Participants with a confirmed or suspected diagnosis of urea cycle disorder (UCD) receiving sodium phenylbutyrate at Baseline.
- Ravicti: Participants with a confirmed or suspected diagnosis of UCD receiving Ravicti at Baseline.
- Sodium Benzoate: Participants with a confirmed or suspected diagnosis of UCD receiving sodium benzoate at Baseline.
- Carglumic Acid: Participants with a confirmed or suspected diagnosis of UCD receiving carglumic acid at Baseline.
- Other: Participants with a confirmed or suspected diagnosis of UCD receiving other (not specified) ammonia-scavenging medication at Baseline.
Period: Overall Study
Arm/Group | Sodium Phenylbutyrate | Ravicti | Sodium Benzoate | Carglumic Acid | Other
Started | 49 | 89 | 4 | 1 | 60
Completed | 42 | 72 | 4 | 1 | 46
Not Completed | 7 | 17 | 0 | 0 | 14
Not completed — Serious Adverse Event | 3 | 0 | 0 | 0 | 1
Not completed — Investigator Request | 0 | 8 | 0 | 0 | 6
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 4
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 1
Not completed — Other, Not Specified | 1 | 9 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Sodium Phenylbutyrate: Participants with a confirmed or suspected diagnosis of UCD receiving sodium phenylbutyrate at Baseline.
- Total: Total of all reporting groups
Arm/Group | Sodium Phenylbutyrate | Ravicti | Sodium Benzoate | Carglumic Acid | Other | Total
Number analyzed (Participants) | 49 | 89 | 4 | 1 | 60 | 203
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.9 (13.5) | 16.7 (15.1) | 9.3 (8.7) | 2.0 (NA) — 1 participant in reporting group | 14.7 (16.9) | 14.5 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 54 | 1 | 0 | 33 | 121
  Male | 16 | 35 | 3 | 1 | 27 | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 16 | 3 | 0 | 7 | 39
  Not Hispanic or Latino | 36 | 73 | 1 | 1 | 53 | 164
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race [Count of Participants; unit: Participants]
  White | 30 | 63 | 4 | 1 | 48 | 146
  Black or African-American | 9 | 9 | 0 | 0 | 4 | 22
  Asian | 1 | 2 | 0 | 0 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 1
  Other, Not Specified | 8 | 15 | 0 | 0 | 5 | 28

OUTCOME MEASURES:

1. Primary Outcome: Mean Blood Ammonia Levels Over Time, by Last Known Ammonia-Scavenging Medication
Description: Retrospective is defined as the 12 months preceding enrollment.
Time Frame: 12 months prior to enrollment (retrospective), Baseline, Day 7 to 30, Month 6, Month 12, Month 18, Month 24, Month 30, Month 36, Month 42, Month 48, Month 54, Month 60, Month 66, Month 72
Population: Participants with a Baseline visit and an assessment at given time point. Participants are grouped by last-known ammonia-scavenging medication at given time point (participants may have been on more than 1 therapy during the study).
Measure: Mean (Standard Deviation); unit: µmol/L
Groups:
- Sodium Phenylbutyrate: Participants with a confirmed or suspected diagnosis of UCD receiving sodium phenylbutyrate.
- Ravicti: Participants with a confirmed or suspected diagnosis of UCD receiving Ravicti.
- Sodium Benzoate: Participants with a confirmed or suspected diagnosis of UCD receiving sodium benzoate.
- Carglumic Acid: Participants with a confirmed or suspected diagnosis of UCD receiving carglumic acid.
- Other: Participants with a confirmed or suspected diagnosis of UCD receiving other (not specified) ammonia-scavenging medication.
Arm/Group | Sodium Phenylbutyrate | Ravicti | Sodium Benzoate | Carglumic Acid | Other
Number analyzed (Participants) | 40 | 67 | 6 | 2 | 5
µmol/L
  Retrospective: number analyzed (Participants) | 19 | 13 | 1 | 1 | 3
  Retrospective | 86.5 (87.13) | 43.8 (27.59) | 23.0 (NA) — 1 participant analyzed | 13.0 (NA) — 1 participant analyzed | 963.7 (721.39)
  Baseline: number analyzed (Participants) | 40 | 67 | 6 | 1 | 0
  Baseline | 64.5 (52.32) | 49.1 (43.58) | 48.0 (29.73) | 21.0 (NA) — 1 participant analyzed |
  Day 7 to 30: number analyzed (Participants) | 7 | 8 | 1 | 0 | 2
  Day 7 to 30 | 64.0 (20.53) | 79.6 (72.23) | 55.0 (NA) — 1 participant analyzed |  | 143.5 (98.29)
  Month 6: number analyzed (Participants) | 28 | 61 | 3 | 2 | 5
  Month 6 | 48.7 (53.77) | 45.0 (30.26) | 190.3 (257.80) | 48.0 (25.46) | 129.4 (110.54)
  Month 12: number analyzed (Participants) | 20 | 60 | 2 | 1 | 2
  Month 12 | 42.4 (20.87) | 39.4 (24.43) | 51.0 (16.97) | 20.0 (NA) — 1 participant analyzed | 79.0 (57.98)
  Month 18: number analyzed (Participants) | 13 | 43 | 3 | 1 | 3
  Month 18 | 54.5 (53.89) | 45.9 (28.26) | 29.0 (11.79) | 13.0 (NA) — 1 participant analyzed | 106.0 (110.31)
  Month 24: number analyzed (Participants) | 13 | 54 | 3 | 1 | 0
  Month 24 | 53.9 (38.49) | 52.8 (78.14) | 43.3 (31.26) | 25.0 (NA) — 1 participant analyzed |
  Month 30: number analyzed (Participants) | 13 | 38 | 4 | 0 | 2
  Month 30 | 42.0 (18.18) | 47.5 (33.27) | 79.8 (85.85) |  | 114.5 (127.99)
  Month 36: number analyzed (Participants) | 10 | 39 | 1 | 0 | 2
  Month 36 | 36.2 (18.90) | 45.9 (34.95) | 72.0 (NA) — 1 participant analyzed |  | 51.5 (34.65)
  Month 42: number analyzed (Participants) | 6 | 32 | 2 | 0 | 0
  Month 42 | 40.2 (14.39) | 43.3 (27.30) | 41.5 (0.71) |  |
  Month 48: number analyzed (Participants) | 7 | 29 | 1 | 0 | 1
  Month 48 | 61.4 (57.78) | 54.2 (42.95) | 36.0 (NA) — 1 participant analyzed |  | 22.0 (NA) — 1 participant analyzed
  Month 54: number analyzed (Participants) | 5 | 15 | 2 | 0 | 1
  Month 54 | 55.6 (8.59) | 45.0 (29.44) | 66.0 (0.00) |  | 292.0 (NA) — 1 participant analyzed
  Month 60: number analyzed (Participants) | 3 | 10 | 1 | 0 | 0
  Month 60 | 57.3 (22.37) | 45.2 (32.78) | 8.9 (NA) — 1 participant analyzed |  |
  Month 66: number analyzed (Participants) | 1 | 4 | 0 | 0 | 0
  Month 66 | 62.0 (NA) — 1 participant analyzed | 31.0 (11.05) |  |  |
  Month 72: number analyzed (Participants) | 1 | 2 | 0 | 0 | 0
  Month 72 | 55.0 (NA) — 1 participant analyzed | 45.5 (43.13) |  |  |

2. Primary Outcome: Median Blood Ammonia Levels Over Time, by Last-Known Ammonia-Scavenging Medication
Description: Retrospective is defined as the 12 months preceding enrollment.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: µmol/L
Arm/Group | Sodium Phenylbutyrate | Ravicti | Sodium Benzoate | Carglumic Acid | Other
Number analyzed (Participants) | 40 | 67 | 6 | 2 | 5
µmol/L
  Retrospective: number analyzed (Participants) | 19 | 13 | 1 | 1 | 3
  Retrospective | 46.0 [18.0 to 304.0] | 38.0 [11.0 to 95.0] | 23.0 [23.0 to 23.0] | 13.0 [13.0 to 13.0] | 1360.0 [131.0 to 1400.0]
  Baseline: number analyzed (Participants) | 40 | 67 | 6 | 2 | 0
  Baseline | 50.0 [12.0 to 247.0] | 37.0 [11.0 to 247.0] | 46.5 [20.0 to 99.0] | 21.0 [21.0 to 21.0] |
  Day 7 to 30: number analyzed (Participants) | 7 | 8 | 1 | 0 | 2
  Day 7 to 30 | 60.0 [32.0 to 93.0] | 61.5 [25.0 to 249.0] | 55.0 [55.0 to 55.0] |  | 143.5 [74.0 to 213.0]
  Month 6: number analyzed (Participants) | 28 | 61 | 3 | 2 | 5
  Month 6 | 33.0 [9.0 to 281.0] | 34.0 [9.0 to 158.0] | 44.0 [39.0 to 488.0] | 48.0 [30.0 to 66.0] | 96.0 [22.0 to 312.0]
  Month 12: number analyzed (Participants) | 20 | 60 | 2 | 1 | 2
  Month 12 | 42.0 [10.0 to 83.0] | 34.5 [9.0 to 122.0] | 51.0 [39.0 to 63.0] | 20.0 [20.0 to 20.0] | 79.0 [38.0 to 120.0]
  Month 18: number analyzed (Participants) | 13 | 43 | 3 | 1 | 3
  Month 18 | 36.0 [20.0 to 226.0] | 45.0 [10.0 to 123.0] | 26.0 [19.0 to 42.0] | 13.0 [13.0 to 13.0] | 51.0 [34.0 to 233.0]
  Month 24: number analyzed (Participants) | 13 | 54 | 3 | 1 | 0
  Month 24 | 47.0 [10.0 to 158.0] | 34.5 [9.0 to 575.0] | 48.0 [10.0 to 72.0] | 25.0 [25.0 to 25.0] |
  Month 30: number analyzed (Participants) | 13 | 38 | 4 | 0 | 2
  Month 30 | 43.0 [19.0 to 81.0] | 35.0 [9.0 to 147.0] | 52.0 [10.0 to 205.0] |  | 114.5 [24.0 to 205.0]
  Month 36: number analyzed (Participants) | 10 | 39 | 1 | 0 | 2
  Month 36 | 38.0 [14.0 to 72.0] | 34.0 [9.0 to 151.0] | 72.0 [72.0 to 72.0] |  | 51.5 [27.0 to 76.0]
  Month 42: number analyzed (Participants) | 6 | 32 | 2 | 0 | 0
  Month 42 | 40.5 [16.0 to 61.0] | 38.0 [10.0 to 124.0] | 41.5 [41.0 to 42.0] |  |
  Month 48: number analyzed (Participants) | 7 | 29 | 1 | 0 | 1
  Month 48 | 39.0 [21.0 to 187.0] | 40.0 [10.0 to 162.0] | 36.0 [36.0 to 36.0] |  | 22.0 [22.0 to 22.0]
  Month 54: number analyzed (Participants) | 5 | 15 | 2 | 0 | 1
  Month 54 | 57.0 [45.0 to 66.0] | 35.8 [12.0 to 134.0] | 66.0 [66.0 to 66.0] |  | 292.0 [292.0 to 292.0]
  Month 60: number analyzed (Participants) | 3 | 10 | 1 | 0 | 0
  Month 60 | 62.0 [33.0 to 77.0] | 29.0 [11.0 to 113.0] | 8.9 [8.9 to 8.9] |  |
  Month 66: number analyzed (Participants) | 1 | 4 | 0 | 0 | 0
  Month 66 | 62.0 [62.0 to 62.0] | 27.5 [22.0 to 47.0] |  |  |
  Month 72: number analyzed (Participants) | 1 | 2 | 0 | 0 | 0
  Month 72 | 55.0 [55.0 to 55.0] | 45.5 [15.0 to 76.0] |  |  |

3. Primary Outcome: Percentage of Participants With Hyperammonemic Crisis (HAC) by Baseline Ammonia-Scavenging Medication, Retrospective Values
Description: Percentage of participants experiencing HAC (reported for the 12 months preceding enrollment).
Time Frame: 12 months prior to enrollment (retrospective)
Population: Participants with a baseline visit.
Measure: Number; unit: percentage of participants
Arm/Group | Sodium Phenylbutyrate | Ravicti | Sodium Benzoate | Carglumic Acid | Other
Number analyzed (Participants) | 49 | 89 | 4 | 1 | 60
percentage of participants | 44.9 | 15.7 | 25.0 | 100.0 | 8.3

4. Primary Outcome: Percentage of Participants With Hyperammonemic Crisis (HAC), Post-Baseline by Last Known Ammonia-Scavenging Medication
Description: Percentage of participants experiencing HAC (post-Baseline).
Time Frame: From enrollment through the end of study (mean overall duration on study was 1187.7 days).
Population: Participants with a baseline visit and at least 1 measurement of this assessment while on therapy. Participants are grouped by last-known ammonia-scavenging medication; participants may have been on more than 1 therapy during the study and the number of participants analyzed may be greater than the overall number of participants.
Measure: Number; unit: percentage of participants
Arm/Group | Sodium Phenylbutyrate | Ravicti | Sodium Benzoate | Carglumic Acid | Other
Number analyzed (Participants) | 61 | 118 | 10 | 2 | 22
percentage of participants | 42.6 | 37.3 | 40.0 | 0 | 72.7

5. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An SAE is an adverse event that: is fatal or life-threatening; results in persistent or significant disability or incapacity. Disability is defined as a substantial disruption of a person's ability to conduct normal life functions; requires inpatient hospitalization or prolongation of an existing hospitalization; is a congenital anomaly/birth defect; any other important medical event that may jeopardize the patient and may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: From enrollment through the end of study (mean overall duration on study was 1187.7 days).
Population: All participants who attended a Baseline visit. Due to data collection complexities in this observational study (e.g., switching of medications, incomplete data on medications, and missing SAE dates) AEs could not be reliably summarized according to a participant's treatment at the time of SAE, and was therefore summarized by treatment at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Phenylbutyrate | Ravicti | Sodium Benzoate | Carglumic Acid | Other
Number analyzed (Participants) | 49 | 89 | 4 | 1 | 60
Participants | 30 | 40 | 2 | 0 | 16

ADVERSE EVENTS:
Time Frame: From enrollment through the end of study (mean overall duration on study was 1187.7 days).
Description: Per protocol, non-serious adverse events were not collected in this observational registry study.
  Due to data collection complexities in this observational study (e.g., switching of medications, incomplete data on medications, and missing SAE dates) AEs could not be reliably summarized according to a participant's treatment at the time of SAE, and was therefore summarized by treatment at baseline.
Arm/Group | Sodium Phenylbutyrate | Ravicti | Sodium Benzoate | Carglumic Acid | Other
All-Cause Mortality (participants affected / at risk) | 3/49 | 2/89 | 0/4 | 0/1 | 1/60
Serious Adverse Events (participants affected / at risk) | 30/49 | 40/89 | 2/4 | 0/1 | 16/60
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sodium Phenylbutyrate (N=49) | Ravicti (N=89) | Sodium Benzoate (N=4) | Carglumic Acid (N=1) | Other (N=60)
Autoimmune Haemolytic Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Immune Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Arginase Deficiency (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0
Eye Swelling (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 3 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 1 | 0 | 0
Diarrhoea Haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Intestinal Perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 7 | 5 | 1 | 0 | 2
Death (General disorders) | 0 | 0 | 0 | 0 | 1
Medical Device Site Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Pneumatosis (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 3 | 2 | 0 | 0 | 0
Bile Duct Stenosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Hepatic Artery Thrombosis (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Anaphylactic Reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Appendicitis Perforated (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Clostridium Difficile Infection (Infections and infestations) | 2 | 0 | 0 | 0 | 1
Corona Virus Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Croup Infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Ear Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Enterobacter Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Escherichia Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 2 | 4 | 0 | 0 | 3
Gastrointestinal Viral Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Human Herpesvirus 6 Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 2 | 2 | 0 | 0 | 2
Medical Device Site Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Metapneumovirus Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Otitis Media Acute (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Pneumonia Respiratory Syncytial Viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Respiratory Syncytial Virus Bronchiolitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Salmonellosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Subcutaneous Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 2
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Viral Infection (Infections and infestations) | 0 | 2 | 0 | 0 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 2 | 1 | 0 | 0 | 0
Accidental Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Procedural Vomiting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0 | 0
Ammonia Increased (Investigations) | 2 | 0 | 0 | 0 | 0
Norovirus Test Positive (Investigations) | 0 | 1 | 0 | 0 | 0
Streptococcus Test Positive (Investigations) | 0 | 1 | 0 | 0 | 0
Transaminases Increased (Investigations) | 0 | 1 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Failure To Thrive (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Feeding Intolerance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Fluid Overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyperammonaemia (Metabolism and nutrition disorders) | 19 | 26 | 0 | 0 | 2
Hyperammonaemic Crisis (Metabolism and nutrition disorders) | 8 | 3 | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Metabolic Disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Altered State Of Consciousness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cerebral Venous Thrombosis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Chorea (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Epileptic Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Febrile Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Guillain-Barre Syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Hyperammonaemic Encephalopathy (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Incoherent (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Ischaemic Stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Metabolic Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Motor Developmental Delay (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 2 | 1 | 0 | 0
Delivery (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0
Device Dislocation (Product Issues) | 1 | 0 | 0 | 0 | 0
Device Occlusion (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Confusional State (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Conversion Disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Mental Status Changes (Psychiatric disorders) | 2 | 3 | 0 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Renal Failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Adnexal Torsion (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Vocal Cord Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Treatment Noncompliance (Social circumstances) | 1 | 0 | 0 | 0 | 0
Spinal Fusion Surgery (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Due to data collection complexities in this observational study (e.g., switching of medications, incomplete data on medications, and missing SAE dates) AEs could not be reliably summarized according to a participant's treatment at the time of SAE, and was therefore summarized by treatment at baseline.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Horizon requests that any investigator/institution that plans on presenting/publishing results provide written notification of their request 60 days prior to their presentation/publication. Horizon requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Horizon needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2013-02-11): https://cdn.clinicaltrials.gov/large-docs/27/NCT01948427/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT01948427/SAP_001.pdf